CLINICAL TRIAL: NCT03579823
Title: Single Centre, Randomised, Single-Blind, Pilot Study to Compare the Safety, Tolerability and Pharmacokinetics of AVT02 to EU-approved Humira® as a Single Dose (40 mg) Subcutaneous Injection in Healthy Adult Subjects (ALVOPAD)
Brief Title: Comparative Safety, Tolerability, Pharmacokinetic Study of AVT02 (100MG/ML) and Humira (100MG/ML) in Healthy Volunteers
Acronym: ALVOPAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVT02-GL-100
Record Dates: First submitted 2018-06-08; First posted 2018-07-09 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Single Centre, Randomised, Single-Blind, Pilot Study
Who Masked: Participant
Masking Description: This study is single blind. Operators are open to treatment allocation. Subjects are blinded to the treatment allocation. In order to keep the blind, subjects are masked during the subcutaneous injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVT02 100 MG/ML (Experimental): Single subcutaneous injection of 40 mg of AVT02 (100MG/ML)
  Interventions: Drug: AVT02 100MG/ML
- Adalimumab 100 MG/ML [HUMIRA] (Active Comparator): Single subcutaneous injection of 40 mg of Adalimumab (100MG/ML) [HUMIRA]
  Interventions: Drug: Adalimumab 100 MG/ML [Humira]

INTERVENTIONS:
Drug: Adalimumab 100 MG/ML [Humira] — prefilled syringe at a concentration of 100MG/ML and delivering 40MG of adalimumab, as a single dose on day 1 day 1
  Arms: Adalimumab 100 MG/ML [HUMIRA]
Drug: AVT02 100MG/ML — prefilled syringe at a concentration of 100MG/ML delivering 40MG of AVT02, as a single dose on day 1 day 1
  Arms: AVT02 100 MG/ML

SUMMARY:
Adalimumab is an immunosuppressive drug that belongs to the family of anti-TNF agents. It contains a monoclonal antibody produced by biotechnology. It is designed to bind to tumor necrosis factor (TNF), a substance that is involved in several auto-immune processes. By binding to TNF, adalimumab blocks its activity, reducing the severity of various chronic inflammatory diseases including Rheumatoid Arthritis, Plaque Psoriasis and others.

Often, the high cost of biologic products may preclude access to the treatment to a big portion of the population worldwide. A biosimilar product that provides comparable safety and efficacy at more affordable cost would fulfill a broader medical need.

Humira has been available on the market for several years. Recently, a higher concentration (100 mg/mL) formulation has been introduced in major markets. Alvotech is developing AVT02, that is a proposed biosimilar of adalimumab containing high concentration (100 mg/mL) of active ingredient.

The objective of this clinical trial is to assess the similarity of AVT02 (100 mg/mL) with Humira (100 mg/mL), in terms of tolerability, safety (including immunogenicity) and compare the pharmacokinetics in healthy volunteers.

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female healthy adult subjects willing to sign an Informed Consent Form and able to undergo protocol related procedures.
* Age: 18 to 55 years, inclusive.
* Body Mass Index (BMI): 19.0 to 30.0 kg per m2.
* Medical history without major pathology, at the discretion of Principal Investigator.
* Resting supine systolic blood pressure of ≤150 mmHg and diastolic blood pressure of ≤90 mmHg. Other vital signs showing no clinically relevant deviations according to the Principal Investigator's judgment.
* Computerised 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the Principal Investigator.
* Subjects who do not smoke tobacco products or use nicotine replacement therapy or e-cigarettes.

Main Exclusion Criteria:

* Evidence of clinically relevant pathology.
* Unable to follow protocol instructions in the opinion of the Principal Investigator.
* History of relevant drug and or food allergies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Known history of previous exposure to adalimumab or other anti-TNF-alpha molecules.
* Any past or concurrent medical conditions potentially increasing the subject's risks, or would have interfered with the study evaluation, procedures, or study completion. Examples of these include medical history with evidence of clinically relevant pathology (e.g., malignancies, demyelinating disorders, herpes zoster, or hepatic, gallbladder or pancreatic diseases).
* Presence of chronic obstructive pulmonary disease. Asthma in the childhood is allowed.
* Evidence of a recent, within 6 months, infection requiring hospitalisation or intravenous antibiotic use.
* Subject has a positive test for Tuberculosis (TB) during screening or a known history of active or latent TB, except documented and complete adequate treatment of TB.
* Having received live vaccines during the 4 weeks before screening or have the intention to receive vaccination during the study.
* Positive for Hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HbcAb), anti- Hepatitis C virus antibodies (HCV), or anti-human immunodeficiency virus (HIV) 1 on 2 antibodies at screening.
* Impaired liver function
* Any persons who are an employee of the Principal Investigator, clinical centre, clinical research organisation or Sponsor, a relative of an employee of the clinical centre, the Investigator, Clinical Research Organization (CRO) or the Sponsor.
* Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline blood pressure at 1, 2, 3, 4, 5, 6, 7, 8, 9, 64 days post dosing | Predose and 1, 2, 3, 4, 5, 6, 7, 8, 9, 64 days post dosing
  Measurement of blood pressure (systolic and diastolic in mm Hg)
Change from baseline heart rate at 1, 2, 3, 4, 5, 6, 7, 8, 9, 64 days post dosing | Predose and 1, 2, 3, 4, 5, 6, 7, 8, 9, 64 days post dosing
  Measure of heart rate (beats per minute)
Change from baseline body temperature at 1, 2, 3, 4, 5, 6, 7, 8, 9, 64 days post dosing | Predose and 1, 2, 3, 4, 5, 6, 7, 8, 9, 64 days post dosing
  Measurement of oral temperature (Celsius degree)
Change from baseline electrocardiogram at 1, 2, 5, 9, 64 days post dosing | Predose and 1, 2, 5, 9, 64 days post dosing
  Analysis of 12-lead electrocardiogram
Change from baseline red blood cells at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure red blood cells count, (unit/mm3)
Change from baseline haemoglobin at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure haemoglobin (g/L)
Change from baseline white blood cells at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure white blood cells count, (unit/mm3)
Change from baseline platelets at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure platelets count, (unit/mm3)
Change from baseline blood gamma glutamyl transferase at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure gamma glutamyl transferase (UI/L)
Change from baseline blood aspartate aminotransferase at 2, 3, 5, 9, 64 days post | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure aspartate aminotransferase (UI/L)
Change from baseline blood alanine aminotransferase at 2, 3, 5, 9, 64 days post | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure alanine aminotransferase (UI/L)
Change from baseline blood potassium at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure potassium (mmol/L)
Change from baseline blood sodium at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure sodium (mmol/L)
Change from baseline blood calcium at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure calcium (mmol/L)
Change from baseline blood phosphate at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure phosphate (mmol/L)
Change from baseline blood chloride at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure chloride (mmol/L)
Change from baseline blood bicarbonate at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure bicarbonate (mmol/L)
Change from baseline blood creatinine at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure creatinine (micromol/L)
Change from baseline blood bilirubin at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure Bilirubin (micromol/L)
Change from baseline international normalised ratio at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure international normalised ratio
Change from baseline prothrombin time at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure prothrombin time (sec)
Change from baseline partial prothrombin time at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure partial prothrombin time (sec)
Change from baseline activated partial thromboplastin time at 2, 3, 5, 9, 64 days post | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure activated partial thromboplastin time (sec)
Change from baseline thrombin time at 2, 3, 5, 9, 64 days post | Predose and 2, 3, 5, 9, 64 days post dosing
  Blood collection to measure thrombin time (sec)
Change from baseline urine leucocytes at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Urine sample collection to measure leucocytes
Change from baseline urine glucose at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Urine sample collection to measure glucose
Change from baseline urine protein at 2, 3, 5, 9, 64 days post dosing | Predose and 2, 3, 5, 9, 64 days post dosing
  Urine sample collection to measure protein

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Over 64 days
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC) of AVT02 and EU Humira
Maximum serum concentration | Over 64 days
  Venous blood samples will be collected for measurement of serum concentration of AVT02 and EU Humira
Time to maximum serum concentration | Over 64 days
  Evaluation of time to maximum plasma concentration (Tmax) of AVT02 and Humira.
Terminal half-life | Over 64 days
  Evaluation of terminal elimination half-life (T1/2) of AVT02 and Humira
Volume of distribution | Over 64 days
  Evaluation of volume of distribution during the elimination phase (Vz) of AVT02 and Humira
Clearance | Over 64 days
  Evaluation of total plasma clearance (CL) of AVT02 and Humira
Incidence and titer of anti-drug antibodies to adalimumab | 15, 29 and 64 days after dosing
  A blood sample will be collected to measure antibodies to AVT02 and Humira

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No